CLINICAL TRIAL: NCT04357314
Title: Myocardial Infarction Rates Overview During COVID-19 Pandemic In France: MODIF Study
Acronym: MODIF
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-03
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Myocardial Infarction
Keywords: Emergency care
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with STEMI in 2019: Patient with acute myocardial infarction between March 17, 2019 and April17, 2019
- Patients with STEMI in 2020: Patient with acute myocardial infarction between March 17, 2020 and April17, 2020.

SUMMARY:
In late December 2019, an emerging disease due to a novel coronavirus (named SARS-CoV-2) rapidly spread in China and outside. France is currently facing the COVID-19 wave with more than 131 863 confirmed cases and almost 25 201 deaths. Systems of care have been reorganized in an effort to preserve hospital bed capacity, resources, and avoid exposure of patients to the hospital environment where COVID-19 may be more prevalent. Therefore, elective procedures of catheterization and programmed hospitalizations have been delayed. However, a significant proportion of procedures within the catheterization laboratory such as ST-elevation myocardial infarction (STEMI), non ST elevation myocardial infarction or unstable angina are mandatory and cannot be postponed. Surprisingly, invasive cardiologist noticed a drop in STEMI volume without reliable data to confirm this impression. Furthermore, a recent single center report in Hong Kong pointed out longer delays of taking care when compared to patients with STEMI treated with percutaneous intervention the previous year. These data are at major concern because delay in seeking care or not seeking care could have detrimental impact on outcomes.

DETAILED DESCRIPTION:
The aim of this study is to investigate the rates and characteristics of patients presenting with acute myocardial infarction between march 1, 2020 to May 31, 2020 and compared those data with those of this year (march 1, 2019 to May 31, 2019).

The following elements will aslo been collected:

* Clinical presentation
* Mode of admission (SAMU (Service d'Aide Médicale Urgente in French ie Emergency Medical Aid Service) / emergency department / in hospital)
* Call for SAMU : delay, number of calls, response
* Thrombolysis
* Delays (symptom onset to first medical contact / door to balloon)
* Final Result : TIMI (Thrombolysis In Myocardial Infarction)
* COVID-19 status if known
* Underlying known ischemic cardiopathy
* ECG (electrocardiogram) Q waves.
* Complication after PCI (Percutaneous Coronary Intervention): Discharged date, LVEF (Left Ventricular Ejection Fraction), ventricular tachycardia Data will be collected through all participating centers under the supervision of the cath lab director.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted on coronary angiography room for acute coronary syndrome with ST segment elevation defined by the following criteria:

* Symptoms suggestive of myocardial ischemia (ex: persistent chest pain) AND
* An elevation of the ST segment (measured from point J) visible on at least two contiguous leads with an elevation ≥ 2.5 millimeters in men <40 years, or ≥ 2 millimeters in men ≥ 40 years, or ≥ 1.5 millimeters in women in V2-V3 leads and / or ≥ 1 millimeter in other leads (in the absence of branch block).

Exclusion Criteria:

- 121/5000

* Contraindication to invasive management related to the general condition of the patient.
* Minors
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the hospital with acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 6332 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a composite of death from all causes and mechanical complications of acute myocardial infarction (MI) | 3 months (between March 1 to May 31, 2019 and between March 1 to May 31, 2020 )
  Free wall rupture, acute ischemic mitral regurgitation, ventricular septal rupture
Rates of patients presenting with acute myocardial infarction | 3 months (between March 1 to May 31, 2019 and between March 1 to May 31, 2020 )
  Compare the number of patients presenting to cardiology department with acute myocardial infarction in 2019 versus in 2020

SECONDARY OUTCOMES:
Patient profile during admission for acute myocardial infarction | 3 months (between March 1 to May 31
  Correlation between clinical patient profile and the degree of affection of regions by COVID-19
Medical care times analysis | 3 months (between March 1 to May 31)
  Correlation between the delay between onset of symptoms - first medical contact - coronary angiography room and the degree of affection of regions by COVID-19
Medical care times analysis | 3 months (between March 1 to May 31, 2019 and between March 1 to May 31, 2020 )
  Delay in minutes from symptom onset and STEMI (ST Segment Elevation Myocardial Infarction) diagnosis; and delay in minutes from onset of symptoms and primary PCI (percutaneous coronary intervention)
Clinical evolution of patients | 3 months (between March 1 to May 31)
  Correlation between the fate of patient and the degree of affection of regions by COVID-19: Number of days in cardiology department, Left Ventricular Ejection Fraction at discharge, presence of hemodynamic complications, presence of mechanical complications, transfer to intensive care unit, infection with COVID-19 during hospitalization, living status at discharge
Clinical evolution of patients | 3 months (between March 1 to May 31, 2019 and between March 1 to May 31, 2020 )
  Number of in hospital outcomes including orotracheal intubation, cardiogenic shock, arrhythmias (ventricular tachycardia of ventricular fibrillation) and in hospital cardiac arrest
STEMI (ST Segment Elevation Myocardial Infarction) admissions incidence rates | 3 months (between March 1 to May 31, 2019 and between March 1 to May 31, 2020 )
  Number of patient admitted in cardiology department with STEMI (ST Segment Elevation Myocardial Infarction)
Proportion of patients who underwent systemic thrombolysis | 3 months (between March 1 to May 31)
  Correlation between the number of patients who underwent systemic thrombolysis and the degree of affection of regions by COVID-19
Proportion of patients infected with COVID-19 | 3 months (between March 1 to May 31)
  Number of patient admitted in cardiology department for acute myocardial infarction infected with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CAYLA, MD, Study Director — Hôpital Universitaire Carémeau; Guillaume BONNET, MD, Principal Investigator — Inserm 970
Locations (1):
- Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No